CLINICAL TRIAL: NCT01514968
Title: A Drug-Drug Interaction Study Between Danoprevir/Low-dose Ritonavir and Cyclosporine, a Potent Inhibitor of OATP, in Healthy Subjects
Brief Title: A Drug-Drug Interaction Study Between Danoprevir/Low-Dose Ritonavir and Cyclosporine in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: NP27947
Record Dates: First submitted 2012-01-16; First posted 2012-01-23 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — Cyclosporine; danoprevir; Ritonavir

ARMS (3):
- DNV/r+cyclosporine (Experimental)
  Interventions: Drug: cyclosporine; Drug: danoprevir; Drug: ritonavir
- cyclosporine (Active Comparator)
  Interventions: Drug: cyclosporine
- danoprevir+ritonavir (Active Comparator)
  Interventions: Drug: danoprevir; Drug: ritonavir

INTERVENTIONS:
Drug: cyclosporine — Single oral dose
  Arms: DNV/r+cyclosporine; cyclosporine
Drug: danoprevir — Single oral dose
  Arms: DNV/r+cyclosporine; danoprevir+ritonavir
Drug: ritonavir — Single oral dose
  Arms: DNV/r+cyclosporine; danoprevir+ritonavir

SUMMARY:
This single-dose, randomized, open-label, 2-sequence, 3-period study will evaluate the effect of cyclosporine on the pharmacokinetics of ritonavir-boosted danoprevir (DNV/r) in healthy volunteers. Subjects will be randomized to one of two treatment sequences to receive a single oral dose of DNV/r or cyclosporine. In treatment period 3, subjects will receive a single oral dose of DNV/r plus cyclosporine. Anticipated time on study is 33 days.

ELIGIBILITY:
Inclusion Criteria:

* Male and female healthy volunteers, 18 to 45 years of age inclusive
* Body mass index (BMI) 18.0 to 32.0 kg/m2
* Weight >/= 50 kg
* Healthy status defined by absence of evidence of any active or chronic disease following detailed medical and surgical history and a complete physical examination
* Nonsmoker
* Females of childbearing potential and males and their female partner(s) of childbearing potential must agree to use 2 forms of contraception, 1 of which must be a barrier method, during the study and for 90 days after the last drug administration (acceptable barrier forms are condom and diaphragm, acceptable non-barrier forms of contraception for this study are non-hormonal intrauterine device and/or spermicide)

Exclusion Criteria:

* Pregnant or lactating females
* Positive results for drugs of abuse in the urine at screening or prior to admission to the clinical site during any study period
* Positive for hepatitis B, hepatitis C or HIV infection
* Current smokers or subjects who have discontinued smoking less than 6 months prior to the first dose of study medication
* Use of hormonal contraceptives (birth control pills, patches or injectable, implantable devices) within 30 days before the first dose of study medication
* Routine chronic use of more than 2 g acetaminophen daily
* Use of any investigational drug or device within 30 days of screening (6 months for biologic therapies) or 5 half-lives of the investigational drug, whichever is longer
* History of clinically significant disease or disorder
* History of clinically significant drug-related allergy (such as anaphylaxis) or hepatotoxicity
* History (within 3 months of screening) of alcohol consumption exceeding 2 standard drinks per day on average (1 standard drink = 10 grams of alcohol)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2011-12; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Effect of single dose of cyclosporine on pharmacokinetics of ritonavir-boosted danoprevir: maximum plasma concentration (Cmax)/area under the concentration-time curve (AUC) | 16 time points up to 96 hours

SECONDARY OUTCOMES:
Effect of single dose of ritonavir-boosted danoprevir on pharmacokinetics of cyclosporine | 16 time points up to 96 hours
Safety: Incidence of adverse events | approximately 50 days

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Lenexa, Kansas, United States

REFERENCES:
- [Derived] Brennan BJ, Moreira SA, Morcos PN, Navarro MT, Asthappan J, Goelzer P, Weigl P, Smith PF. Pharmacokinetics of a three-way drug interaction between danoprevir, ritonavir and the organic anion transporting polypeptide (OATP) inhibitor ciclosporin. Clin Pharmacokinet. 2013 Sep;52(9):805-13. doi: 10.1007/s40262-013-0077-2. PMID 23712757